CLINICAL TRIAL: NCT00189033
Title: Dietary Interventions in Irritable Bowel Syndrome: Soluble, Insoluble or no Fibre? A Randomized Controlled Trial in Primary Care.
Brief Title: Dietary Interventions in Irritable Bowel Syndrome: Soluble, Insoluble or no Fibre?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Maastricht University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJ6Z; 4200.0020
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Colonic Diseases, Functional
Keywords: Irritable Bowel Syndrome; Diet Therapy; Dietary Fiber; Randomized Controlled Trial; Family Practice
MeSH Terms: conditions — Colonic Diseases, Functional; Irritable Bowel Syndrome | interventions — Dietary Supplements; Dietary Fiber

INTERVENTIONS:
Drug: psyllium fibre (dietary supplement)
Drug: wheat bran (dietary supplement)
Drug: rice wheat (placebo)

SUMMARY:
The purpose of this study is to assess the role of dietary fibre in Irritable Bowel Syndrome (IBS) treatment, in particular the role of increasing the content of soluble or insoluble fibres in the daily diet. The primary objective is to compare soluble (psyllium) and insoluble (bran) to placebo, administered over 12 weeks in patients with 'probable' or 'definite' Irritable Bowel Syndrome. The primary efficacy parameter is the responder rate based on weekly assessment of adequate relief of IBS symptoms. Secondary efficacy parameters include changes in IBS related symptoms (abdominal pain, bowel habits) and quality of life.

DETAILED DESCRIPTION:
INTRODUCTION: In daily practice, both patients and doctors consider dietary factors, especially fibre and fluid intake, to play an important role in both the aetiology and the persistence of Irritable Bowel Syndrome (IBS) symptoms. The majority of doctors provides dietary lifestyle advice, targeted at increasing the fibre content of the daily diet by adding insoluble fibre. In addition more than 50% of IBS patients receive pharmacotherapy, frequently including bulking agents, in particular soluble fibres such as psyllium-supplements. There is, however, limited evidence that fibre therapy may alleviate IBS symptoms. In addition, there are indications that insoluble fibres may even worsen IBS symptoms. Scientific evidence pertaining to the different effects of soluble and insoluble fibres on IBS symptoms is very limited indeed, and methodologically sound RCTs in primary care patients are lacking altogether. The latter is important since primary care IBS patients differ in many aspects from secondary/tertiary care patients.

STUDY DESIGN: A double blind parallel-group randomised controlled trial involving IBS patients in primary care comparing 12-week intervention of psyllium fibres, bran, and placebo. After the intervention, all patients will be followed for an additional 12-week period.

STUDY POPULATION: Patients aged 18-65 years presenting to their General Practitioner (GP) with either incident IBS symptoms or with a relapse of pre-existing IBS as well as patients with a prior GP diagnosis of IBS and currently experiencing symptoms are eligible for the study. Patients will be stratified in two equally large patients groups of (a) 'definite' IBS, according to the Rome II diagnostic criteria, and (b) 'probable' IBS, pragmatically diagnosed with IBS by their GP. Patients with alarm symptoms (i.e. abnormalities at physical examination, fever, weight loss, rectal bleeding), with fibre intolerance, with acute abdominal pain, patients with treatment for IBS by a specialist in the prior 48 months, patients with an active psychiatric disorder requiring medication and patients unable to fill out the questionnaires will be excluded.

INTERVENTION: Patients will be randomly allocated to a 12-week treatment period with (a) 10 gram psyllium fibres, (b) 10 gram wheat bran or (c)10 gram identical placebo to be taken in 2 doses with the meal. In healthy subjects, the median intake is 20 gram fibre per day. When focussing on increasing the amount of fibre in the daily diet in IBS treatment, addition of 10 gram fibre to the diet (bringing the total fibre content of the diet to 30 gram), is usually considered adequate. This should be combined with sufficient intake of fluid. All study medication will be filled in comparable pots. To prevent constipation, participants will be instructed not to change dietary habits, and to take an additional 1 litre of fluids daily. Other possible side effects are an unpleasant feeling in de upper gut and rarely allergic reactions such as rash, rhinitis and conjunctivitis. Cellulose can possibly bind glycosides, salicylates, coumarine derivates en nitrofurantoïne. Participants will be instructed to take the fibre at least 2 hours after these medications.

OUTCOME MEASUREMENTS: In line with previous conclusions on optimal outcome assessment in trials on functional GI disease, the primary endpoint is the Adequate Relief question. This measure addresses symptom improvement in IBS treatment with a single question (Did you have adequate relief of IBS-related abdominal pain or discomfort in the past week?) scored on a dichotomous scale. This instrument is a well validated simple outcome assessment for IBS treatment. A positive response is defined as more than 2 weeks Adequate Relief per month. Secondary outcome measures include IBS symptoms, disease specific quality of life, fibre intake, the number of doctor visits, and costs. IBS symptoms will be monitored using the IBS symptom severity score (IBS SSS). This is a well- validated IBS symptom score, which integrates five aspects of bowel dysfunctioning with the actual intensity of IBS symptoms, using visual analogue scales. Disease-specific quality of life will be registrated with the Irritable Bowel Syndrome Quality of Life scale (IBS QOL). This instrument includes 30 items in nine subscales. It has been validated in different populations. Fibre intake will be monitored every 4 weeks using a Food Frequency Questionnaire. Habitual fibre intake can be calculated from the questionnaire data. This instrument is a self-administered food frequency questionnaire and is validated for ranking subjects according to intake for dietary fibre. After the active treatment period of 12 weeks, all patients will be followed up for an additional period of 12 weeks to assess the sustainability of the effects of the interventions. The primary outcome will be measured on a weekly basis. The secondary endpoints will be recorded at 1, 2, 3 and 6 months after start of the intervention, during follow-up visits to the general practitioner. All additional consultations, diagnostics procedures, medication, and referrals during the intervention period will be recorded in the electronic medical file in the practices. Compliance will be checked every visit by the weighting of the contents of the trial medications and registration by a patient's diary.

REQUIRED SAMPLE SIZE: Ninety-five patients are required per treatment arm. Assuming a minimal clinically relevant difference in the proportion of responders (i.e. more than 2 weeks of Adequate Relief per month) between active and placebo treatment of 20%, a placebo response of 40%, a treatment effect of 60% is expected. Taking a type II error of 20% and a type I error of 5% and allowing 10% of dropouts, totally 285 IBS patients are required. Assuming an estimated mean incidence of IBS in primary care, of 8 per 1000 patient years (20 patients per practice per year), an expected inclusion rate of 25%, we expect that 60 general practitioners, each including 5 patients, will be able to include the required number of patients in one year. GPs will be recruited from the Utrecht and Maastricht general practitioners research networks. GPs in both networks have a tradition of participating in academic research and have ample expertise in participating in clinical trials in primary care.

DATA ANALYSIS: Statistical analysis will be based on the intention-to-treat principle. Adequate Relief, IBS Symptom Score and Quality of Life after the 12-week treatment period and after the additional 12-week post-treatment period will be compared with the score at baseline observation (t=0), using Student T-tests for repeated measurements and variance analysis. Stability of the treatment effect in time will be assessed using one-factorial ANOVA for repeated measures. The proportion of responders on the Adequate Relief question (i.e. > 2 weeks Adequate Relief per months) will be compared using chi-square tests. In case of (unexpected) differences in relevant baseline characteristics between the three comparison groups multiple regression analyses will be performed.

ADMINISTRATION: The project will cover 24 months. The first 3 months of the study are necessary to prepare the study. The inclusion period lasts 12 months, 6 additional months are required to complete the follow-up and to perform the first statistical analyses and to prepare the manuscripts. The last 3 months will be used for definitive data analyses and finalisation of the reports.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years presenting to their General Practitioner (GP) with either incident IBS symptoms or with a relapse of pre-existing IBS as well as patients with a prior GP diagnosis of IBS and currently experiencing symptoms are eligible for the study. Patients will be stratified in two equally large patients groups of (a) 'definite' IBS, according to the Rome II diagnostic criteria, and (b) 'probable' IBS, pragmatically diagnosed with IBS by their GP.

Exclusion Criteria:

* Patients treated with fibre in the prior 4 weeks
* Patients with alarm symptoms i.e. abnormalities at physical examination, fever, weight loss, rectal bleeding, acute abdominal pain
* Patient with fibre intolerance
* Patients treated for Irritable Bowel Syndrome by a specialist in the prior 48 months
* Patients with active psychiatric disorder requiring medication
* Patients not able to fill out the questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Adequate Relief of abdominal pain or discomfort.

SECONDARY OUTCOMES:
IBS symptoms (IBS symptom severity score)
IBS related quality of life (IBSQOL)
Fibre intake
The number of doctor visits and costs

CONTACTS AND LOCATIONS:
Overall Officials: Prof. A.W. Hoes, M.D., PhD., Study Chair — UMC Utrecht; C.J. Bijkerk, M.D., Principal Investigator — UMC Utrecht; N.J. de Wit, MD., PhD., Study Director — UMC Utrecht
Locations (2):
- Netherlands (2):
  - University of Maastricht, CAPHRI institute, Department of General Practice, Maastricht
  - University Medical Center Utrecht, Julius Center for Health Sciences and Primary Care, Department of General Practice, Utrecht

REFERENCES:
- [Derived] Bijkerk CJ, de Wit NJ, Muris JW, Whorwell PJ, Knottnerus JA, Hoes AW. Soluble or insoluble fibre in irritable bowel syndrome in primary care? Randomised placebo controlled trial. BMJ. 2009 Aug 27;339:b3154. doi: 10.1136/bmj.b3154. PMID 19713235